CLINICAL TRIAL: NCT04881175
Title: Histological Study to Assess Safety and Efficacy of a Radiofrequency Device Flexible Applicator for Non-Invasive Lipolysis
Brief Title: Histological Study on Safety and Efficacy of a RF Device Flexible Applicator for Non-Invasive Lipolysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was terminated because of a business decision.
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CYN20-FLEX-HISTO
Record Dates: First submitted 2021-05-03; First posted 2021-05-11 (Actual); Results first posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Lipolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- FlexSure Applicator (Experimental): The TempSure FlexSure applicator will be used on the abdomen or flanks.
  Interventions: Device: Non-Invasive Treatment

INTERVENTIONS:
Device: Non-Invasive Treatment — Single-arm group using the FlexSure Applicator device.

SUMMARY:
This is a prospective, open-labeled, non-randomized, multi-center clinical study to collect efficacy data on the TempSure FlexSure applicator for fat lipolysis.

DETAILED DESCRIPTION:
Subjects will attend a screening/pretreatment visit which may be performed on the same day as the treatment visit. Subjects may receive up to 5 treatments every 1-2 weeks on the abdomen or flanks.

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female between the age of 18 - 55 years old.
* Willing to receive treatments with the TempSure device and are willing to have biopsies taken from a control site and the treatment area.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject is currently enrolled in an investigational drug or device trial or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months prior to entering this study.
* The subject has a cut, wound, or infected skin on the area to be treated.
* The subject is on local, oral, or systemic anesthetic agents.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confound study results or may interfere significantly with the subject's participation.
* The subject is currently enrolled in an investigational drug or device trial, or has received an investigational drug or been treated with an investigational device within in the area to be treated 6 months (or at the discretion of the Investigator) prior to entering this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Civiok, Study Director — Cynosure, Inc.
Locations (2):
- United States (2):
  - New Jersey Plastic Surgery, Montclair, New Jersey
  - Bass Plastic Surgery, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gupta V, Sharma VK. Skin typing: Fitzpatrick grading and others. Clin Dermatol. 2019 Sep-Oct;37(5):430-436. doi: 10.1016/j.clindermatol.2019.07.010. Epub 2019 Jul 17. PMID 31896400

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FlexSure Applicator
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | FlexSure Applicator
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 2
  Caucasian | 1
FitzPatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick Skin Score is used to determine skin color. It is a numerical system that classifies skin into six types (Type I, Type II, Type III, Type IV, Type V and Type VI) based on the numerical score achieved (ranging from 0 to 36). The lower the score (and skin type number), the fairer the skin. The higher the score (and skin type number), the more deeply pigmented the skin is. The scale comes from the source listed in the references
  Participants
    Fitzpatrick Skin Type I | 0
    0Fitzpatrick Skin Type II | 0
    Fitzpatrick Skin Type III | 1
    Fitzpatrick Skin Type IV | 0
    Fitzpatrick Skin Type V | 0
    Fitzpatrick Skin Type VI | 2

OUTCOME MEASURES:

1. Primary Outcome: Count of Samples That Showed a Change in Adipocyte Necrosis After Treatment
Description: Photographs of the histological samples before and after the treatment (only one treatment occurred) will be examined for adipocyte necrosis. Each specimen will first be preserved with a fixative and stained with Hematoxylin and eosin (H&E stain). To determine whether or not the samples are expressing histological changes, a pathologist will look at the histology of each individual sample and record if they see any changes in histology post treatment vs. the histology taken at the baseline (these changes are observable to the eye). Then, the number of biopsy samples that express any change in adipocyte necrosis will be reported.
Time Frame: immediately post treatment (only 1 treatment was conducted)
Measure: Number; unit: biopsy samples
Units Other Than Participants: biopsy samples
Arm/Group | FlexSure Applicator
Number analyzed (Participants) | 3
Number analyzed (biopsy samples) | 3
biopsy samples | 0

2. Primary Outcome: Count of Samples That Showed an Inflammatory Immune Response Vs. Baseline
Description: Photographs of the histological samples before and after the last treatment will be examined for an inflammatory immune response. Each specimen will first be preserved with a fixative and stained with Hematoxylin and eosin (H&E stain) To determine whether or not the samples are expressing histological changes, a pathologist will look at the histology of each individual sample and record if they see any changes in histology post treatment vs. the histology taken at the baseline (these changes are observable to the eye). Then, the number of biopsy samples that express any change in an inflammatory immune response will be reported.
Time Frame: Baseline, immediately post treatment (only 1 treatment was conducted)
Measure: Number; unit: biopsy samples
Units Other Than Participants: biopsy samples
Arm/Group | FlexSure Applicator
Number analyzed (Participants) | 3
Number analyzed (biopsy samples) | 3
biopsy samples | 0

ADVERSE EVENTS:
Time Frame: Adverse events were tracked until subject completion of the study, approximately 2 weeks.
Arm/Group | FlexSure Applicator
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FlexSure Applicator (N=3)
skin burn (Skin and subcutaneous tissue disorders) | 2
erythema (Skin and subcutaneous tissue disorders) | 2
pain/tenderness (Skin and subcutaneous tissue disorders) | 2
nodule (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI cannot disclose confidential or proprietary information until after it becomes generally known or available to the public.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT04881175/Prot_SAP_000.pdf